CLINICAL TRIAL: NCT00316784
Title: A Double-Blind, Placebo-Controlled Evaluation of Dose Related Safety and Efficacy of Epicutaneously Applied IDEA-033 for 3 Months Treatment of OA of the Knee Followed by a Double-Blind, Dose-Controlled Evaluation of Safety and Efficacy of Epicutaneously Applied IDEA-033 for 12 Weeks Treatment of OA of the Knee
Brief Title: IDEA-033 Three Months Dose Finding in OA Followed by IDEA-033 Three Months Extension in OA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-033-III-02/E
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis; Knee
Keywords: osteoarthritis; knee; IDEA-033
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

INTERVENTIONS:
Drug: IDEA-033 (and rescue medication)

SUMMARY:
The study objective is the eluciation of the dose-response function in efficacy (and possibly safety) in order to determine an optimal dose with respect to efficacy and safety. The study is designed with three dose levels and one placebo control.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of OA in at least one knee for a minimum of 6 months
* aged 18-75 years old
* eligible subjects must have used an oral or rectal NSAID on at least three days per week during the three months before screening or on at least 25 of the 30 days before screening, but be dissatisfied with the current NSAID treatment
* at baseline visit WOMAC pain subscale at least 40 mm, and at least 15 mm greater than at the screening visit in the index knee
* radiographic evidence consistent with OA criteria of grade 2 or 3 according to Kellgren & Lawrence in the index knee. Radiographs mus have been taken during the 6 months before baseline.
* American College of Rheumatology (ACR) functional class I, II or III

Exclusion Criteria:

* intraarticular injections or arthroscopy of the index knee within 3 months prior to screening, or planned during the study
* history, physical examinations or radiographs suggestive of other rhematic diseases
* known hypersensitivity or contraindication to ketoprofen; NSAID idiosyncrasy
* history of peptic ulcers
* severe liver or gastro-intestinal disease within the last 6 months
* injections or change in oral treatment regimen of glucosamine, chondroitin sulfate, hyaluronic acid, shark cartilage, or vitamin E within 3 months prior to screening
* oral or parenteral corticosteroids within 3 months prior to screening
* analgesic therapy for chronic or recurrent pain conditions for indications other than OA
* immunosuppressants within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704
Dates: Start 2005-07; Study Completion 2006-05

PRIMARY OUTCOMES:
change from baseline at week 12 (or end of study measurements) on the Visual Analogue Scale version of the entire WOMAC Pain subscale (primary)
patient global assessment of response to therapy measured on a 5-point Likert Scale at week 12 or end of study measurements (co-primary)
change from baseline at week 12 (or end of study measurements) on the Visual Analogue Scale version of the entire WOMAC function subscale (co-primary)

SECONDARY OUTCOMES:
Change from baseline at week 12 (or end of study measurements) for Physician's Global Assessment of OA and for observed function (TUG)
Mean number of rescue medication taken per day while in the study
Number of withdrawals and time to discontinuation of the study due to lack of efficacy
Time to onset (in days) of pain relief and time to onset of new flares during treatment
Change from baseline on the vitality subscale of the SF-36 health survey and the EURO QoL

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Stucki, Prof, MD, Principal Investigator — department of physical medicine and rehabilitation of universtity Munich